CLINICAL TRIAL: NCT02187575
Title: Bioequivalence Study of UHAC62XX 10 mg Tablets Compared With 10 mg Capsules Following Multiple Peroral Administration in Healthy Volunteers (An Open-label, Randomised, Two-way Crossover Study)
Brief Title: Bioequivalence Study of UHAC62XX Tablets Compared With Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.259
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- UHAC 62 XX tablet (Experimental)
  Interventions: Drug: UHAC 62 XX tablet
- UHAC 62 XX capsule (Active Comparator)
  Interventions: Drug: UHAC 62 XX capsule

INTERVENTIONS:
Drug: UHAC 62 XX tablet
  Arms: UHAC 62 XX tablet
Drug: UHAC 62 XX capsule
  Arms: UHAC 62 XX capsule

SUMMARY:
Study to investigate the bioequivalence between 10 mg tablets (test drug) and 10 mg capsules (reference drug) of meloxicam (UHAC 62 XX) after 7-day administration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 20 and <= 35 years
* Weight: Body Mass Index >= 18.5 and < 25
* Subjects who are judged by the investigator to be appropriate as the subjects of the study based on results of screening test
* Subjects who volunteer to participate and are able to fully understand and agree with this study by written informed consent

Exclusion Criteria:

* History of gastrointestinal ulcer or surgery of gastrointestinal tract (except appendectomy)
* History of hypersensitivity to UHAC 62 XX and/or salicylate (aspirin etc.) and/or Non-steroidal anti-inflammatory drugs (NSAIDs)
* History of aspirin induced asthma (bronchial asthma induced by NSAIDs)
* History of bleeding tendency
* History of alcohol or drug abuse
* Participation to another trial with an investigational drug within 4 months prior to the trial
* Whole blood donation more than 400 ml within 3 months prior to the trial
* Whole blood donation more than 100 ml within 1 month prior to the trial
* Donation of constituent of blood of more than 400 ml within 1 month prior to the trial
* Any medication which might influence the results of the trial within 10 days prior to the trial
* Excessive physical activities within 7 days prior to the trial
* Alcohol drinking within 3 days prior to the trial
* History of orthostatic hypotension, fainting spells or blackouts
* Other than above, those who are judged by the investigator to be inappropriate as the subjects of the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2002-07; Primary Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration of the analyte in plasma) | up to day 8
AUC 0-τ (Area under the concentration time curve in plasma from zero time to 24 hours after 7-day administration) | up to day 8

SECONDARY OUTCOMES:
Tmax (Time to reach Cmax) | up to day 8
T1/2 (Terminal half-life in plasma) | up to day 8
MRT 0-τ (Mean residence time in the body after 7-day administration) | up to day 8
Cτ (Concentration of the analyte in plasma 24 hours after 7-day administration) | up to day 8
Number of patients with adverse events | up to 20 days after final administration